CLINICAL TRIAL: NCT06958419
Title: Node-Sparing Short-Course Radiotherapy Followed by First-Line Chemotherapy Plus Bevacizumab and PD-1 Inhibitor Versus Chemotherapy Plus Bevacizumab Alone in Metastatic pMMR/MSS Colorectal Cancer: A Randomized, Phase II/III Trial (MODIFI-CRC)
Brief Title: Node-Sparing Short-Course Radiotherapy Plus Chemotherapy, Bevacizumab and PD-1 Inhibitor in Metastatic pMMR/MSS Colorectal Cancer (MODIFI-CRC)
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Yanxin Luo,MD, principle investigator, Sixth Affiliated Hospital, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025ZSLYEC-418
Record Dates: First submitted 2025-04-24; First posted 2025-05-06 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Immune Checkpoint Therapy; Radiotherapy; Metastatic Colorectal Cancer (CRC)
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Node-sparing Radiotherapy Group (Experimental)
  Interventions: Combination Product: Node-Sparing Radiotherapy plus first-line therapy
- First-line therapy Group (Active Comparator)
  Interventions: Combination Product: First-line treatment

INTERVENTIONS:
Combination Product: Node-Sparing Radiotherapy plus first-line therapy — Patients will receive node-sparing modified short-course radiotherapy, followed by 8 cycles of FOLFOX chemotherapy combined with bevacizumab and a PD-1 inhibitor. After induction therapy, patients will continue with maintenance therapy using bevacizumab, PD-1 inhibitor, and 5-fluorouracil (5-FU), administered every 2 weeks (Q2W).
  Arms: Node-sparing Radiotherapy Group
Combination Product: First-line treatment — Patients will receive 8 cycles of FOLFOX chemotherapy combined with bevacizumab, followed by maintenance therapy with bevacizumab and 5-fluorouracil (5-FU), administered every 2 weeks (Q2W).
  Arms: First-line therapy Group

SUMMARY:
The current standard first-line treatment for metastatic colorectal cancer is chemotherapy combined with targeted therapy, yet the prognosis remains poor. Although combining immunotherapy, anti-angiogenic agents, and chemotherapy has shown some efficacy in MSS/pMMR metastatic patients, progression-free survival (PFS) remains suboptimal. Radiotherapy-particularly high-dose radiotherapy-can enhance tumor antigen release and potentially improve the response of MSS/pMMR colorectal cancer to PD-1 inhibitors. Tumor-draining lymph nodes (TDLNs) are key sites for PD-1-mediated anti-tumor activity, but radiation-induced damage and fibrosis may impair their immune function. Prior studies have reported a remarkable pathologic complete response (pCR) rate of 77.8% using node-sparing radiotherapy in locally advanced rectal cancer. This phase II/III study aims to evaluate whether node-sparing modified short-course radiotherapy combined with chemotherapy, bevacizumab, and PD-1 blockade can improve objective response rate (ORR) in phase II and progression-free survival (PFS) in phase III, together with treatment tolerance, and overall prognosis in patients with pMMR/MSS metastatic colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Voluntarily signs a written informed consent form.

  * Aged between 18 and 75 years at the time of enrollment.
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
  * Expected survival of more than 3 months.
  * Histologically or cytologically confirmed colorectal adenocarcinoma.
  * Patients must be considered unsuitable for curative surgical resection or local treatment and must not have received prior systemic anti-tumor therapy for recurrent or metastatic disease. Patients with prior neoadjuvant or adjuvant therapy may be enrolled if recurrence or metastasis occurs ≥12 months after the last dose of such treatment.
  * At least one measurable lesion per RECIST v1.1 that can be accurately measured repeatedly. Note: Brain metastases cannot be used as target lesions.
  * Able to provide 10-20 unstained tumor tissue FFPE slides from recent biopsy or archival material stored within 3 years. Ten slides will be used for immunohistochemistry and ten for genomic testing (recent biopsy preferred). If samples are of insufficient quality (as determined by the central lab), additional slides may be required. If adequate slides cannot be provided, partial or full waiver may be granted upon approval by the medical monitor.
  * Agrees to provide tumor tissue and peripheral blood samples during screening and throughout the study for research purposes.
  * Adequate organ function as defined below:
  * Hematologic (no use of blood products or growth factors within 7 days prior to treatment):
  * Absolute neutrophil count (ANC) ≥ 1.5 × 10⁹/L
  * Platelet count ≥ 100 × 10⁹/L
  * Hemoglobin ≥ 90 g/L
  * Renal:
  * Calculated creatinine clearance (CrCl) ≥ 50 mL/min (Cockcroft-Gault formula: CrCl = [(140 - age) × weight (kg) × 0.85 (if female)] / [72 × serum creatinine (mg/dL)])
  * Urine protein < 2+ on dipstick or < 1.0 g per 24-hour urine collection
  * Hepatic:
  * Total bilirubin (TBil) ≤ 1.5 × upper limit of normal (ULN)
  * AST and ALT ≤ 2.5 × ULN
  * Serum albumin ≥ 28 g/L
  * Coagulation:
  * International normalized ratio (INR) and activated partial thromboplastin time (APTT) ≤ 1.5 × ULN
  * Cardiac:
  * Left ventricular ejection fraction (LVEF) ≥ 50%
  * Women of childbearing potential must have a negative urine or serum pregnancy test within 3 days prior to initiating study treatment. If the urine test is inconclusive, a serum test must confirm the result. Women of childbearing potential engaging in sexual activity with non-sterilized male partners must agree to use acceptable contraception from screening through 120 days after the last dose of study drug. The decision to discontinue contraception beyond this period should be discussed with the investigator. Periodic abstinence and the rhythm method are not acceptable.
  * Women of childbearing potential are defined as those who have not undergone surgical sterilization (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy) and have not been postmenopausal (defined as at least 12 consecutive months of amenorrhea without an alternative medical cause and FSH levels in the postmenopausal range).
  * Highly effective contraception methods are those with a failure rate of <1% per year when used consistently and correctly. In addition to barrier methods, hormonal contraception (e.g., oral contraceptives) must also be used.
  * Willing and able to comply with scheduled visits, treatment procedures, laboratory tests, and other protocol requirements.

Exclusion Criteria:

* • Known MSI-H or dMMR status.

  * History of other malignancies within the past 3 years, except for those cured by local treatment, such as basal cell carcinoma, squamous cell carcinoma of the skin, superficial bladder cancer, or ductal carcinoma in situ of the breast.
  * Prior immunotherapy, including immune checkpoint inhibitors (e.g., anti-PD-1, anti-PD-L1, anti-CTLA-4 antibodies), immune agonists (e.g., ICOS, CD40, CD137, GITR, OX40), or immune cell-based therapies targeting tumor immunity.
  * Prior adjuvant or neoadjuvant therapy targeting EGFR or VEGF/VEGFR pathways (e.g., bevacizumab, cetuximab, panitumumab, aflibercept, regorafenib, or biosimilars).
  * Active CNS metastases. Patients with previously treated brain metastases may be eligible if clinically stable for at least 2 weeks (from the first dose of study drug) and off corticosteroids for at least 3 days prior to treatment. Patients with untreated, asymptomatic brain metastases (no neurologic symptoms, no corticosteroids, and all lesions ≤ 1.5 cm in longest diameter) may enroll but require regular CNS monitoring.
  * Known brainstem, meningeal, or spinal cord metastases or compression.
  * Symptomatic or recurrently drained pleural effusion, pericardial effusion, or ascites.
  * Prior systemic or local anti-tumor therapy for locally advanced rectal cancer, including curative surgery, chemotherapy, radiotherapy, immunotherapy, biologics, or small-molecule targeted therapy.
  * Receipt of nonspecific immunomodulators (e.g., interleukins, interferons, thymic peptides, TNF) within 2 weeks prior to study treatment (except IL-11 for thrombocytopenia), or anti-tumor traditional Chinese medicine within 1 week prior to study treatment.
  * Active autoimmune disease requiring systemic treatment within the past 2 years (e.g., with corticosteroids, immunosuppressants, or DMARDs). Replacement therapy (e.g., thyroid hormone, insulin, or physiologic corticosteroids for adrenal/pituitary insufficiency) is allowed.
  * History of non-infectious pneumonitis requiring systemic corticosteroids, or current interstitial lung disease.
  * History of bleeding disorders or coagulopathy; long-term anticoagulation (e.g., atrial fibrillation with CHADS2 score ≥ 2).
  * Uncontrolled comorbidities including, but not limited to, decompensated cirrhosis, nephrotic syndrome, uncontrolled metabolic disorders, severe active peptic ulcer disease or gastritis, or psychiatric/social conditions impairing protocol compliance or informed consent.
  * History of myocarditis, cardiomyopathy, or malignant arrhythmias; unstable angina, congestive heart failure, or vascular disease (e.g., aortic aneurysm requiring repair or DVT) requiring hospitalization within 12 months. Other cardiovascular conditions affecting drug safety (e.g., poorly controlled arrhythmias, myocardial infarction, or ischemia) are excluded.
  * Within 6 months prior to study treatment: gastroesophageal varices, severe ulcers, unhealed wounds, GI perforation, fistulas, obstruction, intra-abdominal abscess, or acute GI bleeding.
  * Within 6 months prior to treatment: arterial thromboembolism, venous thromboembolism (grade ≥3, NCI-CTCAE v5.0), TIA, stroke, hypertensive crisis, or hypertensive encephalopathy.
  * COPD exacerbation within 1 month before study treatment; uncontrolled hypertension (SBP ≥ 160 mmHg or DBP ≥ 100 mmHg despite oral medications).
  * Active or prior history of inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis, or chronic diarrhea).
  * Serious infections within 4 weeks before treatment, including those requiring hospitalization, sepsis, or severe pneumonia; active infection requiring systemic antibiotics within 10 days before treatment (excluding antiviral therapy for hepatitis B or C).
  * Major surgery or significant trauma within 30 days prior to treatment; minor local surgery within 3 days (excluding PICC line placement).
  * History of immunodeficiency; HIV antibody positivity; long-term use of systemic corticosteroids or immunosuppressants.
  * Known active tuberculosis (TB) or suspected active TB not ruled out by clinical evaluation (e.g., sputum testing, chest imaging); known active syphilis.
  * History of allogeneic organ or hematopoietic stem cell transplantation.
  * Untreated active hepatitis B infection (HBsAg-positive with HBV DNA > 1,000 copies/mL or >200 IU/mL); patients with chronic hepatitis B must receive antiviral therapy during the study. Active hepatitis C (HCV antibody-positive with detectable HCV RNA) is also excluded.
  * Receipt of a live vaccine within 30 days before treatment or planned live vaccination during the study.
  * Known allergy to any component of the study drugs or history of serious hypersensitivity to monoclonal antibodies.
  * Known psychiatric disorders, substance abuse, alcoholism, or drug dependence.
  * Pregnant or breastfeeding women.
  * Any condition, treatment, or laboratory abnormality that may interfere with study results, prevent full participation, or not be in the participant's best interest.
  * Local or systemic disease caused by a benign tumor, or tumor-associated conditions causing high medical risk or survival uncertainty (e.g., leukemoid reaction with WBC > 20 × 10⁹/L, cachexia with >10% weight loss within 3 months prior to screening, or BMI ≤ 18).
  * Current evidence of significant gastrointestinal obstruction based on clinical or radiographic findings.
  * History of bleeding disorders or coagulopathy; radiographic evidence of tumor encasing major vessels or showing necrosis/cavitation that, in the investigator's judgment, may pose bleeding risk; continuous anticoagulation within 10 days prior to first dose.
  * Tumor invasion of critical organs or vessels (e.g., heart/pericardium, trachea, esophagus, aorta, or superior vena cava) with risk of complications such as fistulas (e.g., esophagotracheal, esophageal-pleural, or intestinal fistulas).
  * Presence of free intraperitoneal gas not attributable to recent puncture or local surgical procedure.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) | From initiation of treatment until disease progression or death, whichever occurs first, assessed over a period of up to 36 months
  Phase II: To evaluate whether node-sparing modified short-course radiotherapy combined with chemotherapy, bevacizumab, and a PD-1 inhibitor can improve Objective Response Rate(ORR) in patients with metastatic pMMR/MSS colorectal cancer.
Progression-free survival (PFS) | From initiation of treatment until disease progression or death, whichever occurs first, assessed over a period of up to 36 months
  Phase III: To evaluate whether node-sparing modified short-course radiotherapy combined with chemotherapy, bevacizumab, and a PD-1 inhibitor can improve progression-free survival (PFS) in patients with metastatic pMMR/MSS colorectal cancer.

SECONDARY OUTCOMES:
Duration of response | From the first documented occurrence of complete response (CR) or partial response (PR) to the first documented disease progression (per RECIST v1.1) or death from any cause, whichever occurs first, assessed over a period of up to 36 months
Disease control rate | From treatment start to the end of study at 3 years
Overall survival (OS) rate | From treatment start to the end of study at 3 years
Treatment related adverse effect | From treatment start to 30 days after the end of treatment
Time to response (TTR) | From randomization to the first documented occurrence of complete response (CR) or partial response (PR), assessed over a period of up to 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- The Sixth Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No